CLINICAL TRIAL: NCT07201337
Title: A Randomized, Open-Label, Non-Inferiority Phase III Multicenter Clinical Trial Comparing Reduced-Dose to Standard-Dose Prophylactic Irradiation for Low-Risk Clinical Target Volume (CTV) in the Treatment of Nasopharyngeal Carcinoma.
Brief Title: Reduced-dose vs Standard-dose Irradiation for Low-risk Clinical Target Volume in Nasopharyngeal Carcinoma.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center (Other); First Affiliated Hospital of Guangxi Medical University (Other); Affiliated Hospital of Guangdong Medical University (Other); The University of Hong Kong-Shenzhen Hospital (Other); Dongguan People's Hospital (Other Government); Affiliated Cancer Hospital of Shantou University Medical College (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Principal Investigator, Sun Yet-Sen University Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-FXY-299
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Nasopharyngeal Cancinoma (NPC)
Keywords: Nasopharyngeal Carcinoma; De-escalation; Radiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduced-dose Radiotherapy for Low-risk CTV (Experimental)
  Interventions: Radiation: Radiation Therapy
- Standard-dose Radiotherapy for Low-risk CTV (Active Comparator)
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — PTVnx：70Gy/33Fr；PTVnd：70Gy/33Fr；PTV1：60Gy/33Fr；PTV2：42Gy/26Fr.
  Arms: Reduced-dose Radiotherapy for Low-risk CTV
Radiation: Radiation Therapy — PTVnx：70Gy/33Fr；PTVnd：70Gy/33Fr；PTV1：60Gy/33Fr；PTV2：54Gy/33Fr.
  Arms: Standard-dose Radiotherapy for Low-risk CTV

SUMMARY:
To evaluate the locoregional control, survival rate, toxicity, and quality of life in patients with nasopharyngeal carcinoma treated with reduced prophylactic irradiation doses to the Low-Risk Clinical Target Volume (CTV).

DETAILED DESCRIPTION:
This phase 3, multicenter, non-inferiority, randomized controlled clinical trial recruits patients with newly diagnosed, untreated, non-distant metastatic, non-keratinizing nasopharyngeal carcinoma (NPC). The intervention involves comparing reduced-dose prophylactic irradiation to standard-dose prophylactic irradiation for the low-risk clinical target volume (CTV). The objective is to compare the locoregional control, survival rate, toxicity, and quality of life between the two groups.

ELIGIBILITY:
Inclusion Criteria:

Newly diagnosed, untreated, non-distant metastatic, and non-keratinizing NPC; aged between 18 and 70 years; Eastern Cooperative Oncology Group performance score of 0-1; adequate hematologic function (neutrophil count ≥ 1.5 × 10^9/L, platelet count ≥100×109/L, and hemoglobin≥ 90 g/L); adequate renal function (creatinine ≤ 1.5 upper limit of normal [ULN]) or calculated creatinine clearance (CrCl) ≥ 60 mL/min (Cockcroft-Gault formula); and adequate hepatic function (serum bilirubin ≤ 2.0×ULN, and alanine aminotransferase and aspartate aminotransferase ≤ 2.5×ULN).

Exclusion Criteria:

Previous chemotherapy treatment, surgery (except diagnostic) or radiotherapy to the neck or nasopharyngeal regions; previous malignancy (except for cured basal cell carcinoma or carcinoma in situ of the cervix); lactation or pregnancy; or severe coexisting illness.

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2030-11 (Estimated); Study Completion 2032-11 (Estimated)

PRIMARY OUTCOMES:
Locoregional relapse-free survival | 3 year
  Defined as the time from randomization to either documented local and/or regional relapse or death from any cause (except for metastasis), whichever occurred first.

SECONDARY OUTCOMES:
Overall survival | 3 year
  Defined as the time from randomization to death from any cause.
Failure-free survival | 3 year
  Defined as the time from randomisation to disease recurrence (distant metastasis or locoregional recurrence) or death due to any cause, whichever occurred first.
Distant metastasis-free survival | 3 year
  Defined as the time from randomization to documented distant metastasis or death from any cause (except for locoregional relapse).
Acute toxicities | 3 months
  Occur within 3 months after RT. Acute radiation-related toxicities are assessed using the National Cancer Institute Common Toxicity Criteria version 5.0 scale.
Late toxicities | 3 year
  Occur 3 months after RT, graded according to the Radiation Therapy Oncology Group radiation morbidity scoring criteria
Patient's quality-of-life | 1 year
  Quality-of-life (QoL) scores were assessed using the European Organisation for Research and Treatment of Cancer (EORTC) QoL questionnaire Core 30 items (QLQ-C30) version 3.0 and the head and neck cancer module (QLQ-H and N35).

CONTACTS AND LOCATIONS:
Locations (1):
- Sun yat-sen university cancer center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Huang CL, Zhang N, Jiang W, Xie FY, Pei XQ, Huang SH, Wang XY, Mao YP, Li KP, Liu Q, Li JB, Liang SQ, Qin GJ, Hu WH, Zhou GQ, Ma J, Sun Y, Chen L, Tang LL. Reduced-Volume Irradiation of Uninvolved Neck in Patients With Nasopharyngeal Cancer: Updated Results From an Open-Label, Noninferiority, Multicenter, Randomized Phase III Trial. J Clin Oncol. 2024 Jun 10;42(17):2021-2025. doi: 10.1200/JCO.23.02086. Epub 2024 Mar 20. PMID 38507662
- [Result] Sun XS, Liu SL, Luo MJ, Li XY, Chen QY, Guo SS, Wen YF, Liu LT, Xie HJ, Tang QN, Liang YJ, Yan JJ, Lin DF, Bi MM, Liu Y, Liang YF, Ma J, Tang LQ, Mai HQ. The Association Between the Development of Radiation Therapy, Image Technology, and Chemotherapy, and the Survival of Patients With Nasopharyngeal Carcinoma: A Cohort Study From 1990 to 2012. Int J Radiat Oncol Biol Phys. 2019 Nov 1;105(3):581-590. doi: 10.1016/j.ijrobp.2019.06.2549. Epub 2019 Jul 15. PMID 31319091
- [Result] Tang LL, Huang CL, Zhang N, Jiang W, Wu YS, Huang SH, Mao YP, Liu Q, Li JB, Liang SQ, Qin GJ, Hu WH, Sun Y, Xie FY, Chen L, Zhou GQ, Ma J. Elective upper-neck versus whole-neck irradiation of the uninvolved neck in patients with nasopharyngeal carcinoma: an open-label, non-inferiority, multicentre, randomised phase 3 trial. Lancet Oncol. 2022 Apr;23(4):479-490. doi: 10.1016/S1470-2045(22)00058-4. Epub 2022 Feb 28. PMID 35240053
- [Result] Mao YP, Wang SX, Gao TS, Zhang N, Liang XY, Xie FY, Zhang Y, Zhou GQ, Guo R, Luo WJ, Li YJ, Liang SQ, Lin L, Li WF, Liu X, Xu C, Chen YP, Lv JW, Huang SH, Liu LZ, Li JB, Tang LL, Chen L, Sun Y, Ma J. Medial retropharyngeal nodal region sparing radiotherapy versus standard radiotherapy in patients with nasopharyngeal carcinoma: open label, non-inferiority, multicentre, randomised, phase 3 trial. BMJ. 2023 Feb 6;380:e072133. doi: 10.1136/bmj-2022-072133. PMID 36746459
- [Result] Tang LL, Chen L, Xu GQ, Zhang N, Huang CL, Li WF, Mao YP, Zhou GQ, Lei F, Chen LS, Huang SH, Chen L, Chen YP, Zhang Y, Liu X, Xu C, Zhao Y, Li JB, Liu N, Xie FY, Guo R, Sun Y, Ma J. Reduced-volume radiotherapy versus conventional-volume radiotherapy after induction chemotherapy in nasopharyngeal carcinoma: An open-label, noninferiority, multicenter, randomized phase 3 trial. CA Cancer J Clin. 2025 May-Jun;75(3):203-215. doi: 10.3322/caac.21881. Epub 2025 Feb 19. PMID 39970442